CLINICAL TRIAL: NCT07140627
Title: COMPARISON OF BUPIVACAINE WITH AND WITHOUT DEXMEDETOMIDINE IN CAUDAL BLOCK AMONG CHILDREN UNDERGOING INGUINAL HERNIOTOMY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allama Iqbal Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 65
Record Dates: First submitted 2025-08-22; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pain; Rescue Analgesia
Keywords: Bupivacaine; Dexmedetomidine; Inguinal herniotomy; Rescue Analgesia
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A with 0.25% Bupivacaine only (Experimental): After ethical approval, patients who met inclusion criteria were enrolled after obtaining written consent from their parents. Using computer-related random numbers, patients were allocated in two groups of 30: Group A Included 30 participants and received Bupivacaine alone. A 22G cannula was used to perform a caudal block in the left lateral position under sterile conditions following the induction of anesthesia and before the surgery. The attending physician recorded postoperative pain every two hours using the Wong-Baker Faces Pain Scale. Intravenous Paracetamol (10 mg/kg/dose) was given as rescue analgesia if the patient reported a pain score of ≥4, and the duration of the administration was recorded. Structured proforma were used to record all pertinent data.
  Interventions: Drug: Bupivacain
- Group B with 0.25% Bupivacaine and Dexmedetomidine (Experimental): After ethical approval, patients who met inclusion criteria were enrolled after obtaining written consent from their parents. Using computer-related random numbers, patients were allocated in two groups of 30: Group B Included 30 participants and received Bupivacaine alone. A 22G cannula was used to perform a caudal block in the left lateral position under sterile conditions following the induction of anesthesia and before the surgery. The attending physician recorded postoperative pain every two hours using the Wong-Baker Faces Pain Scale. Intravenous Paracetamol (10 mg/kg/dose) was given as rescue analgesia if the patient reported a pain score of ≥4, and the duration of the administration was recorded. Structured proforma were used to record all pertinent data.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.

INTERVENTIONS:
Drug: Bupivacain — A 22G cannula was used to perform a caudal block in the left lateral position under sterile conditions following the induction of anesthesia and before the surgery. 30 participants had received 1 mL/kg 0.25% bupivacaine. Post operative pain was assessed.
  Arms: Group A with 0.25% Bupivacaine only
Drug: Dexmedetomidine & Bupivacaine. — A 22G cannula was used to perform a caudal block in the left lateral position under sterile conditions following the induction of anesthesia and before the surgery. 30 participants were included and administered 1 mL/kg 0.25% bupivacaine and 1 μg/kg dexmedetomidine. Post operative pain was assessed.
  Arms: Group B with 0.25% Bupivacaine and Dexmedetomidine

SUMMARY:
A random controlled trial, was held at Jinnah Hospital in Lahore, consisting of 60 male pediatrics (6 months to 12 years), who were undergoing unilateral inguinal herniotomy or hydrocele repair. Patients were randomly allocated in two groups: Group A alone received 1 mL/kg 0.25% bupivacaine, while Group B received the same dose with 1 μg/kg dexmedetomidine. The pain score was evaluated by Wong-Beker Face Scale postoperatively every two hours, rescue analgesia (intravenous paracetamol 10 mg/kg) when the pain score reached ≥4

ELIGIBILITY:
Inclusion Criteria:

* Male children who were undergoing elective unilateral inguinal herniotomy or hydrocele surgery

Exclusion Criteria:

* Patients were excluded if they were already on analgesic (according to medical records)
* Obstructed inguinal hernias or bilateral hernias (confirmed through ultrasound)

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | 2 hourly assessment for 8 hours on basis of pain score
  In both groups the attending physician recorded postoperative pain every two hours using the Wong-Baker Faces Pain Scale. Intravenous Paracetamol (10 mg/kg/dose) was given as rescue analgesia if the patient reported a pain score of ≥4, and the duration of the administration was recorded. Structured proforma were used to record all pertinent data.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Muhammad Umer Iqbal Butt, MBBS FCPS, Principal Investigator — Allama Iqbal Medical College/Jinnah Hospital Lahore
Locations (1):
- Allama Iqbal Medical College/ Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No